CLINICAL TRIAL: NCT01265212
Title: Prevalence of Human Papillomavirus in Men Living in the Northern Plains
Status: Completed | Type: Observational
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Other Study IDs: IISP ID: 37392
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Epithelial skin swabs collected for the purpose of HPV DNA detection. DNA extraction and HPV testing will be performed.
Oversight: Data Monitoring Committee: No

SUMMARY:
HPV infection is associated with cervical and other anogenital cancers. HPV may also be associated with the development of prostate cancer. The purpose of the study is to determine the prevalence of HPV infection in men living in South Dakota.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ages 18-65
* Living in South Dakota (AKA Northern Plains)

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male residents of South Dakota.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of HPV in men living on the Northern Plains | No time point

CONTACTS AND LOCATIONS:
Overall Officials: Diane Maher, PhD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Health, Sioux Falls, South Dakota, United States